CLINICAL TRIAL: NCT02856906
Title: An Follow-up Study of Occlusal Adjustment for Orofacial Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meiqing Wang (Other)
Responsible Party: Sponsor-Investigator, Meiqing Wang, Professor, State Key Laboratory of Military Stomatology, Department of Oral Anatomy and Physiology, School of Stomatology, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Department of Oral Anatomy
Record Dates: First submitted 2016-07-15; First posted 2016-08-05 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Orofacial Pain; Trigeminal Neuralgia
Keywords: Orofacial Pain; Electromyography; dental occlusion
MeSH Terms: conditions — Facial Pain; Trigeminal Neuralgia; Bites and Stings | interventions — Occlusal Adjustment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Occlusal adjustment group (Experimental): Patients in this group will receive treatment of occlusal adjustment based on the clinical and lab examination results.
  Interventions: Other: occlusal adjustment

INTERVENTIONS:
Other: occlusal adjustment

SUMMARY:
The purpose of this study is to determine whether what kind of occlusion are related the orofacial pain under investigation, and whether occlusal adjustment have an effect in relief of this kind of orofacial pain.

DETAILED DESCRIPTION:
1. T-scan analysis system is used to record the occlusal contact relationships. And at same time, Electromyographic recording system is used to record the Masseter (MM) and Anterior Temporalis (TA) muscles' surface electromyographic (SEMG) in the two time points: before the treatment and 4-weeks follow-up after treatment.

   After recording, several parameters is taken to indicate the occlusal changes when researchers set the T-Scan occlusal parameters as 100% intercuspal position (ICP) maximum voluntary clenching (MVC), 75% ICP-MVC, 50% ICP-MVC, 25% ICP-MVC, and the number of occlusal contact and the values of the the Masseter (MM) and Anterior Temporalis (TA) muscles' surface electromyographic (SEMG) values is acquired by the software in the screen.
2. Occlusal imprints which indicates the their occlusal relationships is made by researchers when the volunteers ICP clenching in the two time points: before the treatment and 4-weeks follow-up after treatment.

   Break-over and the sub-break-over point of the occlusal imprints is amplified by software. The investigators compute the number and area about that.
3. The investigators also recorded frequency of attack and score of visual analogue scale (VAS), the dosage of drug, and short form-McGill-2 in the follow-ups time frame: immediately after the first treatment, 1-, 4-, 12- and 24-weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patients claim orofacial pain. The pain has been treated but not relieved by medication, surgery, root canal therapy, even teeth extracting, or the pain relieve effect went down for a period. The patients also match the following item 1 or 2:
* Item 1: disorder characterized by recurrent unilateral brief electric shock-like pains, abrupt in onset and termination, limited to the distribution of one or more divisions of the trigeminal nerve and triggered by innocuous stimuli. It may develop without apparent cause or be a result of another diagnosed disorder. There may or may not be, additionally, persistent background facial pain of moderate intensity.They fulfilled criteria A-E
* At least three attacks of unilateral facial pain fulfilling criteria B and C
* Occurring in one or more divisions of the trigeminal nerve, with no radiation beyond the trigeminal distribution
* Pain has at least three of the following four characteristics:

  * recurring in paroxysmal attacks lasting from a fraction of a second to 2 minutes.
  * severe intensity.
  * electric shock-like, shooting, stabbing or sharp in quality.
  * precipitated by innocuous stimuli to the affected side of the face.
* No clinically evident neurological deficit
* Not better accounted for by another the International Classification of Headache Disorders 3rd edition diagnosis.
* Item 2 Persistent facial and/or oral pain, with varying presentations but recurring daily for more than 2 hours per day over more than 3 months, in the absence of clinical neurological deficit.They fulfilled criteria A-E
* Facial and/or oral pain fulfilling criteria B and C
* Recurring daily for >2 hours per day for >3 months
* Pain has both of the following characteristics: 1. poorly localized, and not following the distribution of a peripheral nerve 2. Dull, aching or nagging quality
* Clinical neurological examination is normal
* A dental cause has been excluded by appropriate investigations
* Not better accounted for by another the International Classification of Headache Disorders 3rd edition diagnosis

Exclusion Criteria:

* Head and facial trauma; orofacial and/or intracranial space occupying lesion indicated by craniofacial CT ; pain caused by sinusitis and acute pulpitis, periapical periodontitis and periodontitis disease; no occlusal abnormalities and occlusion treatment indications through a series of occlusal examination; children (younger than 18 years old) and pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain reduction assessed on the Visual Analog Scale（VAS） | 4-weeks after the treatment

SECONDARY OUTCOMES:
Pain reduction assessed on the Visual Analog Scale（VAS） | 1-, 12-, 24-weeks after the treatment
Attack frequency | 1-,4-,12-,24-weeks after the treatment
  Times of attack per day stand for attack frequency
Pain reduction assessed on the short form-McGill-2 | 1-,4-,12-,24-weeks after the treatment
  Pain' levels reduction assessed on score of short form-McGill-2 .
The dosage of medicine | 1-, 4-, 12-, 24-weeks after the treatment.
  Grams per day of patients take the medicine .

OTHER OUTCOMES:
Number of break-over point of occlusal imprints. | 4-weeks after treatment
Number of sub-break-over point of occlusal imprints. | 4-weeks after treatment
Area of break-over point of occlusal imprints(cm2) . | 4-weeks after treatment
  Area of break-over point of occlusal imprints(cm2) is computed by software.
Area of sub-break-over point of occlusal imprints(cm2). | 4-weeks after treatment
  Area of sub-break-over point of occlusal imprints(cm2) is computed by software.
Occlusal force ratio（%）in position (ICP)- maximum voluntary clenching (MVC). | 4-weeks after the treatment
  The T-scan analysis system indicates the value of left and right side occlusal force ratio（%）in position (ICP)- maximum voluntary clenching (MVC).
Number of occlusal contact in T-Scan system in ICP-MVC | 4-weeks after the treatment
  The T-scan analysis system indicates the number of left and right side occlusal contact in ICP-MVC.
Anterior Temporalis (TA) muscles' surface electromyographic(SEMG)（uV) in ICP-MVC. | 4-weeks after the treatment
  The system indicates left and right side Anterior Temporalis (TA) muscles' surface electromyographic(SEMG) （uV）in ICP-MVC.
Masseter (MM) surface electromyographic(SEMG)（uV）in ICP-MVC. | 4-weeks after the treatment
  The system indicates right and left side Masseter (MM) surface electromyographic(SEMG)（uV）in ICP-MVC.
Occlusal force ratio（%）of dental arch in lateral cuspal to cuspal. | 4-weeks after treatment
  T-scan analysis system indicates the value of working and non-working side dental arch occlusal force ratio（%) in lateral cuspal to cuspal.
Number of occlusal contact in lateral cuspal to cuspal | 4-weeks after treatment
  T-scan analysis system indicates number of occlusal contact of working and non-working side in lateral cuspal to cuspal.
Anterior Temporalis (TA) muscles' surface electromyographic(SEMG)（uV） in lateral cuspal to cuspal. | 4-weeks after treatment
  The system indicates working and non-working side Anterior Temporalis (TA) muscles' surface electromyographic(SEMG)（uV）in lateral cuspal to cuspal.
Masseter (MM) surface electromyographic(SEMG)（uV）in lateral cuspal to cuspal. | 4-weeks after treatment
  The system indicates non-working and working side Masseter (MM) surface electromyographic(SEMG)（uV）in lateral cuspal to cuspal.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoxiong Guo, M.D, Study Chair — State Key Laboratory of Military Stomatology, Department of Oral Anatomy and Physiology and TMD，School of Stomatology, The Fourth Military Medical University, Xi 'an, China.
Locations (1):
- State Key Laboratory of Military Stomatology, Department of Oral Anatomy and Physiology and TMD，School of Stomatology, The Fourth Military Medical University, Xi 'an, China., Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No